CLINICAL TRIAL: NCT00802191
Title: WiiMote Game Controller as a Device to Study Movement Disorders
Status: Terminated | Type: Observational
Why Stopped: Lack of study participants, no data published.
Sponsor: Vanderbilt University (Other)
Collaborators: National Parkinson Foundation (Other); Robertson County Parkinson Support Group (Unknown)
Responsible Party: Principal Investigator, Thomas L Davis, MD, Vanderbilt University
Other Study IDs: TDavis Wii
Record Dates: First submitted 2008-12-02; First posted 2008-12-04 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Parkinson Disease; Essential Tremor
MeSH Terms: conditions — Parkinson Disease; Essential Tremor

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control Group: Participants with no movement disorders.
- Movement Disorders Participants: Participants have a movement disorder

SUMMARY:
Purpose of the study:

The purpose of this study is to investigate the Wii remote game control device for use in the study of Movement Disorders. The term "Movement Disorders" refers to a group of abnormal medical conditions characterized by involuntary body movements. Current treatment of these disorders is primarily geared to improve symptoms. Rating scales are usually used to grade response to treatment. These rating scales require special training, take a lot of time, and often present with great variability. Thus, the development of a simple device to perform efficacy measurements offers a great advantage over current methods and is less costly.

DETAILED DESCRIPTION:
The expected length of taking part in this study will depend on whether or not subjects are chosen for a group to look at the reproducibility of the data collected from the Wii remote. If subjects agree to take part in the study, basic data including age, gender, ethnicity, and medications will be collected. If subjects have been diagnosed with a movement disorder, that diagnosis will also be recorded. This data will be secured in a HIPAA compliant computer system and recorded data will be given a unique random code. During the Wii remote portion of the study, subjects will be asked to hold the Wii remote controller in several different positions and perform various movements with the controller.

These include:

1. Holding the controller still with the elbow straight and then the elbow bent.
2. Tapping the control button as fast as you can.
3. Rotation of your wrist as fast as you can.
4. Bending at the wrist and at the elbow as fast as you can.
5. Walking 30 feet.
6. Attaching the controller to your arm with a Velcro strap and repeating the motions performed while holding the controller.

These maneuvers will be done first with the right and then the left hand. We expect that this series will take about 5 minutes.

If subjects have Parkinson's disease they will also be asked to undergo Part III (Motor Sub-Scale) of the Unified Parkinson's Disease Rating Scale. This scale measures various aspects such as finger tapping, hand opening and closing and walking on a scale of 0 - 4. We expect that this portion of the examination will take about 5 minutes.

If subjects carry the diagnosis of Essential Tremor, they will be asked to undergo Standard Measure of EssentialTremor that includes drawing of spirals and pouring of water from one glass to another. Again, we estimate that this scale will take about 5 minutes.

If subjects carry the diagnosis of Parkinson's disease or Essential Tremor and have deep brain stimulation surgery, results of using the Wii™ Remote game controller (handheld or attached using a Velcro strap) will be done during a clinical programming appointment. The information obtained will not be used for any clinical use and will not interfere with the normal standard of care.

A sub-set of patients will be asked to repeat these measures at various times to see if there is either a learning curve, or if the measures are repeatable over time. Subjects may decline this at any point in time.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, aged 18 or older, with abnormal movements (including tremor, chorea, dystonia, myoclonus, and tic) and normal controls (subjects without abnormal movements).
2. Subjects must be willing and able to comply with study procedures.
3. Patients must be willing and able to give meaningful, written informed consent.

Exclusion Criteria:

1. Significant cognitive impairment which, in the opinion of the Investigator, would interfere with the ability to complete all the tests required in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 18 Years and older, females of childbearing potential, healthy volunteers and adults with movement disorders.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2007-08; Primary Completion 2013-05 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas L Davis, MD, Principal Investigator — Department of Neurology/Movement Disorders
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States